CLINICAL TRIAL: NCT04851015
Title: Low Dose Trimethoprim-Sulfamethoxazole for the Treatment of Pneumocystis Jirovecii Pneumonia
Acronym: LOW-TMP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Todd C. Lee MD MPH FIDSA, Associate Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-7386
Record Dates: First submitted 2021-04-12; First posted 2021-04-20 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Pneumocystis; Pneumocystis Pneumonia; Pneumocystis Jirovecii Infection; Pneumocystis Infections; Pneumocystis Carinii Infection; Pneumocystosis; Pneumonia (Etiology); Pneumocystis Carinii; Infection, Resulting From HIV Disease; Pneumocystosis Associated With AIDS
Keywords: Pneumocystis; PCP; PJP
MeSH Terms: conditions — Pneumonia, Pneumocystis; Pneumocystis Infections; Pneumonia; Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Off-Label Use

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced dose TMP-SMX (Experimental): Trimethoprim-Sulfamethoxazole at a total dose of 10mg/kg/day. Oral or intravenous drug will be administered at discretion of treating team. This will be given as a dose of 10mg/kg/day open label with additional placebo tablets or intravenous placebo solution given to simulate 15mg/kg/day. All doses will be adjusted for obesity and renal function.
  Interventions: Drug: trimethoprim-sulfamethoxazole
- Standard dose TMP-SMX (Active Comparator): Trimethoprim-Sulfamethoxazole at a total dose of 15mg/kg/day. Oral or intravenous drug will be administered at discretion of treating team. This will be given as 10mg/kg/day open label plus an extra masked 5mg/kg/day of tablets or intravenous solution. All doses will be adjusted for obesity and renal function.
  Interventions: Drug: trimethoprim-sulfamethoxazole

INTERVENTIONS:
Drug: trimethoprim-sulfamethoxazole — 10mg/kg/day of TMP component
  Other Names: Reduced dose
  Arms: Reduced dose TMP-SMX
Drug: trimethoprim-sulfamethoxazole — 15mg/kg/day of TMP component
  Other Names: Standard dose
  Arms: Standard dose TMP-SMX

SUMMARY:
Pneumocystis jirovecii pneumonia (PJP) is an opportunistic fungal infection of immunocompromised hosts which causes in significant morbidity and mortality. The current standard of care, trimethoprim-sulfamethoxazole (TMP-SMX) at a dose of 15-20 mg/kg/day of TMP, is associated with serious adverse events, including hypersensitivity reactions, drug-induced liver injury, cytopenia, and renal failure occurring among 20-60% of patients. The frequency of adverse events increases in a dose dependent manner and commonly limits the use of TMP-SMX.

Reduced treatment doses of TMP-SMX for PJP reduced ADEs without mortality differences in a recent meta-analysis of observational studies. We therefore propose a Phase III randomized, placebo-controlled trial to directly compare the efficacy and safety of low dose (10 mg/kg/day of TMP) compared to the standard-of-care (15 mg/kg/day) among patients with PJP for the primary outcome of death, new mechanical ventilation, and change of treatment.

DETAILED DESCRIPTION:
Pneumocystis jirovecii pneumonia (PJP) is an opportunistic fungal infection primarily affecting immunocompromised patients. Adults with HIV (particularly CD4 ≤200 cells/µL), solid organ and allogeneic hematopoietic stem cell transplant recipients, as well as patients on certain chemotherapies, immunosuppressant drugs, and systemic corticosteroids are at a highest risk. Although routine primary prophylaxis has diminished its prevalence, PJP still results in significant morbidity and mortality worldwide. Retrospective cohort studies have reported mortality rates between 20-50% among non-HIV populations and 10-20% for patients with HIV.

Current guidelines from the National Institutes of Health (NIH), the HIV Medicine Association of the Infectious Diseases Society of America (IDSA), and the American Society of Transplantation (AST) all recommend weight-based trimethoprim-sulfamethoxazole (TMP-SMX) at a dose of 15-20 mg/kg/day of the trimethoprim component as the standard of care. Yet, higher doses of TMP-SMX are associated with serious adverse events, including hypersensitivity reactions, drug-induced liver injury, cytopenia, and renal failure with adverse drug events (ADEs) reported among 20-60% of patients on treatment.

To better inform the optimal dosing strategy for PJP therapy, we recently performed a systematic review and meta-analysis of reduced dose regimens of TMP-SMX in the treatment of PJP among immunocompromised adult patients with and without HIV. When comparing standard doses to reduced doses (≤10mg/kg/day of the TMP component), there was no statistically significant difference in mortality (absolute risk difference: -9% in favor of reduced dose, 95% CI: -27% to 8%) with a corresponding 18% (95% CI: -31% to -5%) absolute risk reduction of Grade III or higher adverse events. These data provide the best available evidence for treatment equipoise and highlight the need for a randomized controlled trial to directly compare dosing strategies.

The primary objective of this trial is to determine whether treatment with reduced-dose TMP-SMX (10mg/kg/day) is superior to standard dose (15mg/kg/day) among immunocompromised HIV-infected and uninfected patients with PJP for the composite primary outcome of death, new mechanical ventilation, or change in treatment by Day 21.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised (including but not limited to HIV, solid organ transplant, solid tumors, hematological stem cell transplant and malignancies, systemic diseases, chemotherapy, long term corticosteroid use, and immunosuppressive therapies, as well as primary immunodeficiencies
* Presentation to a day hospital, emergency department, or admitted to hospital
* Proven or probable diagnosis of PJP using an adapted version of the 2021 EORTC/MSGERC criteria.

Exclusion Criteria:

* Previous severe adverse reaction to TMP-SMX, any sulfa drug, or any component of formulation
* Compliant with PJP prophylaxis for ≥4 weeks with TMP-SMX at enrollment
* More than 72 hours of any therapy for PJP
* Hepatic impairment marked by alanine aminotransferase levels ≥5 times the upper limit of normal
* Known G6PD deficiency
* Known diagnosis of porphyria
* Known pregnancy or breastfeeding (as per Health Canada)
* Unable to provide informed consent and no available healthcare proxy (with ethics approval for deferred consent in cases of critical illness); refusal of consent; no reliable means of outpatient contact (telephone/email/text);
* Previously enrolled

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Proportion with Treatment failure | 21 days
  Composite of death, new mechanical ventilation or treatment change for presumed inefficacy or severe adverse events

SECONDARY OUTCOMES:
Proportion who die | 21 days
  All cause mortality
Proportion who require new mechanical ventilation | 21 days
  A new requirement for mechanical ventilation
Proportion with treatment change due to inefficacy | 21 days
  Treatment change for presumed inefficacy
Proportion with treatment change due to toxicity | 21 days
  Treatment change for drug toxicity
Proportion with ongoing oxygen need | Day 7
  Requirement for oxygen according to guidelines for oxygen use in hospitalized patients
Proportion with ongoing oxygen need | Day 14
  Requirement for oxygen according to guidelines for oxygen use in hospitalized patients
Proportion with ongoing oxygen need | Day 21
  Requirement for oxygen according to guidelines for oxygen use in hospitalized patients
Proportion requiring new non-invasive ventilation | 21 days
  New non-invasive ventilation (e.g. BiPAP, high-flow nasal canulae)
Proportion with new renal failure | 21 days
  New grade 3 or 4 renal failure by Common Terminology Criteria for Adverse Events definition and by modified KDIGO: increase in serum creatinine by≳26.5 umol/l within 48 hours; or increase in serum creatinine to ≳1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or new hemodialysis, wherein hemodialysis was not previously required.
Proportion with hyperkalemia | 21 days
  Proportion with Grade 3 or 4 hyperkalemia (non-hemolyzed sample) by Common Terminology Criteria for Adverse Events definition
Proportion with drug-induced hepatitis | 21 days
  Proportion with Grade 3 or 4 drug-induced hepatitis by Common Terminology Criteria for Adverse Events definition
Proportion with Skin rash | 21 days
  Proportion with development of a Grade 3 or 4 skin rash (by Common Terminology Criteria for Adverse Events definition) that was intolerable to the patient, persisted unabated for 48 hours or more, or had bullae or mucous-membrane involvement.
Proportion with new cytopenias | 21 days
  Proportion with development of new Grade 3 or 4 cytopenias by Common Terminology Criteria for Adverse Events definition
Proportion with hypoglycemia | 21 days
  Proportion with greater than 3 episodes of documented capillary or blood hypoglycemia (≤2.5mmol/L)
EQ-5D-5L | Day 28
  Quality of life as measured by EQ-5D-5L and interpreted based on Canadian value set (see Med Care. 2016 Jan;54(1):98-105)
Quality of life measured by visual analog scale | Day 28
  Measured by VAS for quality of life (higher is better from 0-100)

OTHER OUTCOMES:
Proportion with all cause mortality | 90 days
  All cause mortality
Proportion with at least 1 recurrence of Pneumocystis | 90 days
  A subsequent diagnosis of pneumocystis pneumonia occurring between days 22 and 90

CONTACTS AND LOCATIONS:
Overall Officials: Emily G McDonald, MD MSc, Principal Investigator — Research Institute of the McGill University Health Centre; Todd C Lee, MD MPH FIDSA, Principal Investigator — Research Institute of the McGill University Health Centre; Zahra N Sohani, MD PhD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre (Royal Victoria Hospital and Montreal General Hospital), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
A copy of a trial data required to replicate trial publication analyses will be shared within 3-6 months of publication.
  After study completion, a fully de-identified copy of the full trial dataset can be made available to other researchers subject to a data sharing agreement enacted under Quebec law.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 3-6 months post publication
Access Criteria: Trial data and analytic code required to replicate any analyses presented in the publication will be shared openly via a website which we will set up at that time.
  For a copy of the complete de-identified dataset, we will require a formal data sharing agreement (enacted under Quebec law) between the requesting group and the RI-MUHC.

REFERENCES:
- [Background] Butler-Laporte G, Smyth E, Amar-Zifkin A, Cheng MP, McDonald EG, Lee TC. Low-Dose TMP-SMX in the Treatment of Pneumocystis jirovecii Pneumonia: A Systematic Review and Meta-analysis. Open Forum Infect Dis. 2020 Apr 2;7(5):ofaa112. doi: 10.1093/ofid/ofaa112. eCollection 2020 May. PMID 32391402
- [Derived] Sohani ZN, Butler-Laporte G, Aw A, Belga S, Benedetti A, Carignan A, Cheng MP, Coburn B, Costiniuk CT, Ezer N, Gregson D, Johnson A, Khwaja K, Lawandi A, Leung V, Lother S, MacFadden D, McGuinty M, Parkes L, Qureshi S, Roy V, Rush B, Schwartz I, So M, Somayaji R, Tan D, Trinh E, Lee TC, McDonald EG. Low-dose trimethoprim-sulfamethoxazole for the treatment of Pneumocystis jirovecii pneumonia (LOW-TMP): protocol for a phase III randomised, placebo-controlled, dose-comparison trial. BMJ Open. 2022 Jul 21;12(7):e053039. doi: 10.1136/bmjopen-2021-053039. PMID 35863836